CLINICAL TRIAL: NCT00797095
Title: Health Behaviors in School-Age Children: 2009/2010
Brief Title: Health Behaviors in School-age Children: 2009-2010
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909023; 09-CH-N023
Record Dates: First submitted 2008-11-22; First posted 2008-11-25 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2014-10-20

CONDITIONS: Obesity; Substance Abuse; Violence; Mental Health
Keywords: Adolescence; Obesity; Substance use; Prevalence; Social and Environmental Contexts; Survey
MeSH Terms: conditions — Obesity; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The Health Behaviors in School-age Children (HBSC) study is a consortium of investigators from 40 predominantly European and North American countries who conduct a common survey of early adolescent health behaviors every 4 years. The survey gathers information about nutrition, dieting practices, physical activity, injuries, violence, relationships with family and friends, perceptions of school as a supportive environment, alcohol and tobacco use and drug use among adolescents, and about the communities in which students live. The U.S. sponsors of the survey are the National Institutes of Health and the Health Resources and Services Administration. This is the fourth survey done in the United States.

The objectives of the international HBSC study are:

* To assess the prevalence of early adolescent health behaviors
* To identify psychosocial factors associated with adolescent behaviors
* To provide an opportunity for analyses of cross-national comparisons
* To provide an opportunity for analyses of trends in the U.S. and cross-nationally

In addition to the above, the survey includes additional questions designed to provide information about areas of specific national interest, including the following:

* To assess the association of school, family, peers, and other environmental factors on health behavior and health status
* To assess the prevalence and identify factors associated with obesity, diet and physical activity
* To assess the prevalence and identify factors associated with bullying and risk behaviors.

This is the fourth U.S. administration of the HBSC survey, previously administered in 1997-1998, 2001-2002, and 2005-2006.

About 16,000 students in grades 5 thorough 10 at randomly selected public and private schools across the United States complete a 30- 40-minute survey. The questionnaires are anonymous; students are instructed not to put their name on the survey. When they finish the survey, they place it in an envelope and seal it. The envelopes are then put in a box. Reports do not include the names of participating counties, cities, school districts, schools, or students.

The information collected from U.S. school children is compared with similar information collected from school children in 40 other countries. The survey is used to help set national priorities for school and youth programs, as well as to monitor the progress of these programs.

DETAILED DESCRIPTION:
The Health Behaviors in School-age Children (HBSC) survey is the only international survey of its type that includes a national survey of adolescent health behavior in the U.S. The U.S. HBSC complements the Youth Risk Behavior Survey (YRBS) and the Monitoring the Future surveys of older adolescents. The aims of the survey are to assess the prevalence of health behaviors and identify contextual factors associated with them in a national probability sample of 6th to 10th grade students, allowing for trend analyses and cross-national comparisons among the 40 countries involved in the quadrennial international HBSC surveys. This would be the fourth U.S. administration of the HBSC survey, previously administered in 1997/1998, 2001/2002, and 2005/2006. Because core survey items have remained consistent both nationally and internationally since 2001, the 2009/2010 survey would provide essential data for examining national and international trends.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any children in the randomly selected classrooms being surveyed who have active or passive parental consent (depending on the requirements of the particular school district and school).

EXCLUSION CRITERIA:

- Special education classrooms will not be surveyed.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12651 (Actual)
Dates: Start 2008-11-19; Study Completion 2014-10-20

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Simons-Morton, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brener ND, Kann L, Kinchen SA, Grunbaum JA, Whalen L, Eaton D, Hawkins J, Ross JG. Methodology of the youth risk behavior surveillance system. MMWR Recomm Rep. 2004 Sep 24;53(RR-12):1-13. PMID 15385915
- [Background] Eaton DK, Brener ND, Kann L, Pittman V. High school student responses to different question formats assessing race/ethnicity. J Adolesc Health. 2007 Nov;41(5):488-94. doi: 10.1016/j.jadohealth.2007.05.017. Epub 2007 Aug 29. PMID 17950169
- [Background] Johnston LD, Delva J, O'Malley PM. Sports participation and physical education in American secondary schools: current levels and racial/ethnic and socioeconomic disparities. Am J Prev Med. 2007 Oct;33(4 Suppl):S195-208. doi: 10.1016/j.amepre.2007.07.015. PMID 17884568